CLINICAL TRIAL: NCT05070806
Title: Plastic Surgery Training in Europe
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Other Study IDs: 21/06/099
Record Dates: First submitted 2021-09-20; First posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Plastic Surgery Training

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Survey study to evaluate plastic surgery training in European countries.

DETAILED DESCRIPTION:
National delegates of 30 European countries - the 27 member countries of the European Union (Austria, Belgium, Bulgaria, Croatia, Cyprus, Czech Republic, Denmark, Estonia, Finland, France, Germany, Greece, Hungary, Ireland, Italy, Latvia, Lithuania, Luxembourg, Malta, The Netherlands, Poland, Portugal, Romania, Slovakia, Spain and Sweden) and Norway, Switzerland and the United Kingdom were invited to complete a questionnaire on plastic surgery training.

ELIGIBILITY:
Inclusion Criteria:

* Countries of the European Union (Austria, Belgium, Bulgaria, Croatia, Cyprus, Czech Republic, Denmark, Estonia, Finland, France, Germany, Greece, Hungary, Ireland, Italy, Latvia, Lithuania, Luxembourg, Malta, The Netherlands, Poland, Portugal, Romania, Slovakia, Spain and Sweden) and Norway, Switzerland and the United Kingdom
* Countries must organise plastic surgery training

Exclusion Criteria:

* Countries other than member states of the European Union, Norway, Switzerland and United Kingdom
* Countries that do not provide plastic surgery training

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Twenty-seven member countries of the European Union (Austria, Belgium, Bulgaria, Croatia, Cyprus, Czech Republic, Denmark, Estonia, Finland, France, Germany, Greece, Hungary, Ireland, Italy, Latvia, Lithuania, Luxembourg, Malta, The Netherlands, Poland, Portugal, Romania, Slovakia, Spain and Sweden) and Norway, Switzerland and the United Kingdom
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Organisation of training | 2019-2020
  Organisation of training (e.g. centralised or decentralised, number of training centres, number of trainees, etc)
Scope of practical training curriculum | 2019-2020
  Scope of practical training curriculum (e.g. number of clinical rotations, number of surgical procedures, types of surgical procedures, etc)
Scope of theoretical courses | 2019-2020
  Scope of theoretical courses (e.g. topics that are included in theoretical courses, hours of theoretical courses, etc)
Evaluation of trainees | 2019-2020
  Evaluation of trainees (e.g. number of oral examinations, number of MCQ examinations, number of written examinations, etc)

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Belgium